CLINICAL TRIAL: NCT04281238
Title: The Effects of Yoga Training in Ankylosing Spondylitis Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of Covid-19
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Yasemin ACAR, Research assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/07-20
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Ankylosing Spondylitis; Yoga
Keywords: ankylosing spondylitis; yoga
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga group (Experimental): Participants in this group will be given yoga training 3 days a week for 8 weeks. In addition, patients in this group will be taught home exercises and asked to do these exercises 5 days a week for 8 weeks.
  Interventions: Other: Yoga group
- Control group (Other): Patients in this group will be taught home exercises and asked to do these exercises 5 days a week for 8 weeks.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Yoga group — Yoga training 3 days a week for 8 weeks. In addition to this, home exercises 5 days a week for 8 weeks
  Arms: yoga group
Other: Control group — Home exercises 5 days a week for 8 weeks
  Arms: Control group

SUMMARY:
The aim of the study is to investigate the effect of yoga training on functional level, disease activity, spinal mobility, balance, sleep quality, depression and quality of life in AS patients.

DETAILED DESCRIPTION:
Yoga is an ancient Indian practice, dating back several thousand years, with objective of uniting mind, body, and spirit. In Western cultures, Hatha yoga is most commonly practiced, and generally includes a set of physical poses(asanas), breathing techniques(pranayama) and deep relaxation(savasana).Yoga has been shown to increase mobility, reduce pain, and improve quality of life in many diseases. However, there is no study examining the effects of yoga training in AS patients.Therefore, the aim of this study is to investigate the effects of yoga training in AS patients.

60 AS patients aged 20-60 years will be randomly assigned to yoga or control group. Home exercises will be taught to both groups, and a brochure with home exercises will be given. The yoga group will participate in a yoga class 3 days a week, during 8 weeks. The control group will not participate in a yoga class, only will do home exercises. Assessments will be done at baseline and after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ankylosing spondylitis(AS) patients diagnosed according to modified New York criteria
* To be volunteer

Exclusion Criteria:

* the presence of peripheral enthesitis, orthopedic disorders, cardiovascular disorders, neurological disorders, visual and auditory deficits,
* history of surgery for spine or lower limb,
* failure to complete the test

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Spinal Metrology Index (BASMI) | 5 minutes
  Asses spinal mobility. The total score ranges from 0 to 10. Higher scores mean poor spinal mobility.

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 2 minutes
  Assess disease activity. The total score ranges from 0 to 10. High scores mean an increase in disease activity.
Bath Ankylosing Spondylitis Functional Index (BASFI) | 3 minutes
  Assess functional capacity. This self-assessment instrument consists of eight specific questions regarding function in AS and two questions reflecting the patient's ability to cope with everyday life regarding function in AS and two questions reflecting the patient's ability to cope with everyday life.The BASFI score is calculated by dividing the sum of the scores from 10 questions by 10.
Short Form-36 (SF-36) | 6 minutes
  Assess quality of life
Beck Depression Inventory | 5 minutes
  Assess depression
Beck Anxiety Inventory | 4 minutes
  Assess anxiety
Pittsburgh Sleep Quality Index | 4 minutes
  Assess quality of sleep
Balance Master system | 10 minutes
  Assess balance

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül University, Izmir, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided